CLINICAL TRIAL: NCT05079165
Title: EVALUATION OF THE RESPONSE TO mRNA SARS-CoV-2 VACCINE IN A COHORT OF LIVER TRANSPLANTED OR LISTED PATIENTS
Brief Title: Covid Vaccination in Liver Transplantation
Acronym: VACCHEPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8261
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Coronavirus Vaccine; COVID-19 Pandemic; COVID-19 Virus Disease; SARS-CoV-2 Infection; Solid organ transplant; mRNA vaccine; MODERNA; liver transplant; Serological testing; serological response; SARS-CoV-2 mRNA vaccine; Anti-SARS-CoV-2 IgG antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective study is to evaluate the proportion of seroconversion after 2 doses mRNA anti-SARS-CoV2 vaccination in a cohort of high risk liver transplanted patients.

Seroprevalence is a secondary objective in order to identify seronegative patients with a history of COVID-19 (ie who lost antibodies) and seropositive patients with no history of COVID-19.

The hypothesis is that the degree of immunosuppression is determinant on the seroconversion rate and therefore, although at higher risk of severe forms of COVID-19, liver transplanted patients have a lower chance of being protected after vaccination.

Seroconversion rate in previously seronegative and with no history of COVID-19 liver transplanted patients is the main evaluation criteria.

The factors associated with the absence of seroconversion will be identified as a potential tool to better adapt the vaccination strategy in this population.

The rate of seroconversion after the 1st dose will also be evaluated. Safety of the 1st and 2nd injection will be reported as well as their value to predict seroconversion.

A control group of patients listed for transplantation will also be included both in the seroprevalence and the seroconversion analysis.

Persistance of the antibodies in long-term after transplantation and after transplantation for the patients who have been vaccinated before transplantation will also be reported.

ELIGIBILITY:
Inclusion criteria:

* Liver transplanted patients for > 6 months after transplantation
* Listed cirrhotic patients
* Age >18 years-old
* Consent for vaccination with mRNA vaccine

Exclusion criteria:

* Vaccination with non mRNA anti-SARS-CoV-2 vaccine
* Expressed opposition to participation to the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Liver transplanted adult patients for > 6 months after transplantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the serological response to the anti-SARS-CoV-2 mRNA vaccine | Files analysed retrospectively from January 18, 2020 to April 30, 2021 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service deChirurgie Générale Hépatique-Endocrinienne,et transplantation - Hôpitaux Universitaires de Strasbourg, Strasbourg, France